CLINICAL TRIAL: NCT00387556
Title: Does Ondansetron Reduce the Incidence of Vomiting When Used in Conjunction With Ketamine During Procedural Sedation in the Pediatric Emergency Department
Brief Title: Ondansetron Reduce Vomiting Associated With Ketamine PSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02-0528
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Conscious Sedation
Keywords: ketamine; children; emesis
MeSH Terms: conditions — Vomiting | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine + Ondansetron (Experimental): ketamine 1 mg/kg IV (maximum single dose 100 mg)+ondansetron (0.15 mg/kg/dose; maximum dose 4 mg)
  Interventions: Drug: Ondansetron
- Ketamine + Placebo (Placebo Comparator): ketamine 1 mg/kg IV (maximum single dose 100 mg)+2 ml normal saline solution IV (placebo
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Drug: Ondansetron — ondansetron (0.15 mg/kg/dose; maximum dose 4 mg)
  Other Names: Zofran

SUMMARY:
Ondansetron, a commonly used anti-vomiting medication, may reduce the occurrence of vomiting associated with ketamine during procedural sedation in the pediatric emergency department.

ELIGIBILITY:
Inclusion Criteria:

* age 1-21 years, ASA I or II, fracture of dislocation reduction

Exclusion Criteria:

* age < 1 year, ASA III or IV, hypertension, glaucoma, acute globe injury, increased intracranial pressure or central nervous system mass lesion, major psychiatric disorder, porphyria, previous adverse reaction to ketamine or ondansetron, parent, guardian or patient unwilling to provide informed consent.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 268 (Actual)
Dates: Start 2002-12; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
incidence of vomiting | Duration of ED stay and after discharge
  The primary outcomes in this study were vomiting in the ED and after discharge, as determined by telephone follow-up

SECONDARY OUTCOMES:
Length of ED stay | Duration of ED stay
  Secondary outcome measures were length of ED stay
Satisfaction with Sedation | Length of ED stay.
  patient or parent satisfaction with their sedation

CONTACTS AND LOCATIONS:
Overall Officials: Joe E Wathen, MD, Principal Investigator — University of Colorado Health Science Center
Locations (1):
- The Childrens Hospital, Denver, Colorado, United States